CLINICAL TRIAL: NCT06383767
Title: A Open-label, Randomized, Multicenter Phase III Study of ESG401 Versus Investigator's Choice Chemotherapy in Patients With Locally Advanced or Metastatic HR+/HER2- Breast Cancer Who Had Failed at Least One Line of Chemotherapy
Brief Title: A Phase III Study of ESG401 for Locally Advanced or Metastatic HR+/HER2- Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESG401-301
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Capecitabine; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESG401 for injection (Experimental): IV infusion on day 1, 8 and15 of each 28 day cycle
  Interventions: Drug: ESG401
- Treatment of Physician's Choice (Active Comparator): Eribulin 1.4 mg/m2, IV infusion on day 1 and 8 of each 21 day cycle
  Capecitabine 1000 or 1250 mg/m2, po, from day 1 to 14 of each 21 day cycle
  Vinorelbine 25 mg/m2, IV infusion on day 1 and 8 of each 21 day cycle
  Gemcitabine 1000 mg/m2, IV infusion on day 1,8 and 15 of each 28day cycle
  Interventions: Drug: Eribulin, capecitabine, gemcitabine or vinorelbine (Treatment of Physician's Choice)

INTERVENTIONS:
Drug: ESG401 — IV infusion on day 1,8, and 15 of each 28 day cycle
  Arms: ESG401 for injection
Drug: Eribulin, capecitabine, gemcitabine or vinorelbine (Treatment of Physician's Choice) — Eribulin, capecitabine, gemcitabine or vinorelbine
  Arms: Treatment of Physician's Choice

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of ESG401 in patients with unresectable locally advanced or metastatic HR+/HER2- breast cancer.

DETAILED DESCRIPTION:
This is a open-label, randomized, multicenter Phase 3 study to evaluate ESG401 versus Treatment of Physician's Choice (TPC) in subjects with unresectable locally advanced or metastatic HR+/HER2- breast cancer who had failed at least one line of systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals able to understand and give written informed consent.
* Males or females aged ≥ 18 years ;
* Histologically and/or cytologically confirmed HR+/HER2- breast cancer who had failed at least one line of systemic chemotherapy in metastatic settings;
* Patients who are eligible for a chemotherapy regimen in the control group;
* Patients with at least one measurable lesion per RECIST 1.1 criteria;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1;
* Expected survival ≥ 12 weeks;
* Patients with adequate organ and bone marrow function;
* Female patients of childbearing potential and male patients with partners of childbearing potential who use effective medical contraception from the time of signing the informed consent form until 180 days after the last dose.

Exclusion Criteria:

* Received chemotherapy, targeted therapy, immunotherapy, interventional therapy or other systemic anti-cancer therapie within 4 weeks before the first investigational product administration;
* Toxicities from prior anti-tumor therapy not recovering to ≤ Grade 1;
* Received major surgeries 4 weeks prior to the first dose of study treatment or planned to receive major surgeries during the study ;
* Prior topoisomerase I inhibitor therapy, including antibody-drugconjugate(ADC) therapy, or prior TROP2 targeted therapy, or use of any investigational anti-cancer drug within 28 days or 5 half-lives before the first investigational product administration;
* New thromboembolic events, intestinal obstruction, gastrointestinal bleeding or perforation within 6 months;
* Uncontrolled systemic bacterial, viral or fungal infections;
* Subjects with symptomatic or untreated CNS metastases, or those requiring ongoing treatment for CNS metastases;
* Patients with Primary CNS malignancy；or patients with other malignancies within 3 years prior to the first dose;
* Patients with uncontrollable systemic diseases;
* Patients with gastrointestinal diseases (such as chronic gastritis, chronic enteritis or gastric ulcers), or with a previous history of severe or chronic diarrhea;
* Subjects with clinically significant cardiovascular disease;
* Human Immunodeficiency Virus (HIV) infection;
* Active hepatitis B or hepatitis C;
* Known immediate or delayed hypersensitivity reaction to irinotecan or other camptocampin derivatives such as topotecan or to have had grade ≥3 gastrointestinal reactions associated with irinotecan, or allergies, or to any investigational drug or excipient ingredient;
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by IRC per RECIST 1.1 | Up to 24 months
  PFS was defined as the time from randomization to PD or death, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free survival (PFS) assessed by the investigators per RECIST V 1.1 | Up to 24 months
  PFS was defined as the time from randomization to PD or death, whichever occurs first.
Overall Survival (OS) | Up to 24 months
  OS was defined as the time from randomization to death.
Objective Response Rate (ORR) | Up to 24 months
  ORR was defined as the proportion of of patients with a CR and PR assessed by IRC and investigators per RECIST v 1.1
Clinical Benefit Rate (CBR) | Up to 24 months
  CBR was defined as the proportion of patients with a CR or PR or with SD at Week 24 assessed by IRC and investigators per RECIST v 1.1
Duration of Response (DoR) | Up to 24 months
  From the date that response criteria are first met to the first occurrence of PD as determined by BIRC and investigators per RECIST v1.1 or death from any cause, whichever occurs first.
Quality of life evaluated using the NCC-BC-A scale | Up to 24 months
  To assess the impact of ESG401 on disease related symptoms and quality of life of patients using the NCC-BC-A scale
Adverse events(AEs) and severe adverse events (SAEs) | From signing the ICF up to last dose plus 30 days
  Incidence and severity of AEs and SAEs (per CTCAE 5.0), and clinically significant abnormal laboratory findings
Clearance | Up to 24 months
  Mean population clearance will be derived from pooled data of drug concentrations. Covariates of influence on drug clearance will be incorporated within a population pharmacokinetic model.
Volume of distribution | Up to 24 months
  Mean population volume of distribution will be derived from pooled data of drug concentrations. Covariates of influence on volume of distribution will be incorporated within a population pharmacokinetic model.
ADA | Up to 24 months
  Incidence of anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No